CLINICAL TRIAL: NCT01709396
Title: Extended Dose - Total Body Irradiation Followed By Allogeneic Stem Cell Transplantation For The Treatment Of Refractory Acute Leukemia And Advanced Myelodysplastic Syndrome
Brief Title: ED-TBI Followed By Allogeneic Stem Cell Transplantation For The Treatment Of Refractory AML And Advanced MDS
Acronym: ED-TBI
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: initial on hold due to space but now permanently suspended due to futility.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011064-01
Record Dates: First submitted 2012-10-12; First posted 2012-10-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Acute Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18 cGY ED-TBI (Experimental): 18 cGY ED-TBI followed by an allogenic done marrow transplant
  Interventions: Radiation: ED-TBI

INTERVENTIONS:
Radiation: ED-TBI — Patients will receive 18Gy ED-TBI in 8 fractions of 2.25 Gy each, twice/day for 4 days. Following the final fraction of TBI and an allogeneic hematopoietic stem cell graft.

SUMMARY:
Acute myeloid leukemia (AML) is a rapidly fatal malignancy of the bone marrow. It can be treated with chemotherapy alone, in some cases, but in the majority of cases, the only treatment that can cure the disease is an allogeneic stem cell transplant, with a cure rate of 30-40%. In another subset, the disease is less responsive to chemotherapy and in these aggressive forms, its cure rate is no better than 20% beyond 2 years, and is usually rapidly fatal within 6 months.

Therefore, for this most aggressive form of the disease, modifications to the transplant protocol are required in order to try to improve on these poor results. There are a number of areas within the transplant protocol on which modifications can be made in order to achieve these goals. These include: higher doses of chemotherapy and or radiation; alterations of the new bone marrow graft; and alterations of the immune suppression, enhancing the graft vs. leukemia effect. By focusing on one or more of these components, one might be able to enhance the anti-leukemic aspect of the treatment resulting in a more successful outcome.

One aspect the investigators, in Ottawa, have focused on is the initial intensive conditioning regimen, specifically the radiation component. It is the investigators belief that in the most resistant disease it is important to use the highest tolerable anti-leukemic treatment upfront, specifically, enhancing the radiation component of the initial conditioning regimen. Previous studies have suggested that higher doses of radiation might be more effective at eliminating the disease, however, toxicity and logistics of delivering the radiation have limited its use. Technical advances in the delivery of radiation have now permitted the safer use of high doses of radiation.

Through modifications to the transplant procedure, the investigators believe that they can deliver higher doses of radiation safely and this will translate into improved outcomes in this high-risk subgroup of patients with AML.

Study Objectives

The goal of this study is to determine if a total dose of 18Gy ED-TBI followed by an alloHSCT for patients with refractory AML will result in an improved progression-free survival.

DETAILED DESCRIPTION:
Study Rationale

1. AML is a bone marrow based malignancy that is rapidly growing and rapidly fatal if left untreated. Despite therapeutic strategies for up to 70% of patients, 20% are primarily refractory and another 50% will relapse after first line therapy. Among these refractory and relapsed patients the only, potentially, effective therapy is an alloHSCT, however, long-term survival rates range from as low as <10% up to 20%.
2. Increased doses of radiation in the form of TBI to a threshold of 15.75 Gy with chemotherapy have been demonstrated to reduce the relapse rate significantly; however, OS is compromised by the high rate of toxicity.
3. Evidence suggests that escalated doses of radiation are possible, which offers the potential to increase the dose of radiation to as much as 20Gy, safely.
4. Locally, increased doses of radiation without chemotherapy did not demonstrate any significant toxicity up to a dose of 16Gy.
5. Therefore, as proposed a radiation-only stem cell transplant would allow us to test the hypothesis that increased doses of radiation will reduce the relapse rate while minimizing the toxicity in a very high-risk population of patients with AML, resulting in an improved progression-free and overall survival.

Trial Design

This is a single institution, Phase II study examining the efficacy and toxicity of ED-TBI followed by an alloHSCT on patients with high risk, refractory acute myeloid leukemia.

Treatment Overview

Patients who have met the inclusion criteria will receive a myeloablative dose of radiation followed by an alloHSCT. Acute radiation and transplant related toxicity will be evaluated as the maximum value on the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v.4), during the first 30 days following the transplantation and the LENT-SOMA Radiation Toxicity Scale. The radiation dose to the lungs and kidneys as well as the total dose received by the other organs will be considered independently for the purposes of determining the maximum tolerated radiation dose for that body region.

Eligibility Assessments

Assessments to determine the eligibility to participate in this study will be performed before enrollment in the study, but after the subject has signed the informed consent. Subjects who do not meet the eligibility criteria will be considered screening failures and will not be enrolled.

These assessments will determine:

* Subject eligibility for entry on study,
* Suitability to undergo TBI followed by an alloHSCT.
* Pre-treatment leukemia activity.

The following pre-treatment assessments will be performed within a six-week period prior to enrollment:

* History and physical examination, including height, weight, vital signs
* ECOG Performance Status and Karnofsky performance status (appendix #3).
* CBC, differential, platelets, and reticulocyte count.
* INR, PTT, fibrinogen
* Serum electrolytes, urea, creatinine, calcium and phosphorus, AST, ALT, ALP, total bilirubin and LD
* Pre-transplant infectious disease markers:CMV serology, HIV-1 and HIV-2, HTLV-1 and HTLV-2, HBsAg, Anti-HBs, Anti-HBc, Anti-HCV, Serologic Test for Syphilis (STS)
* Electrocardiogram (ECG).
* Echocardiogram including measurement of LVEF.
* Pulmonary function tests including FEV1, FVC and DLCO.
* Pregnancy test (urine or serum βHCG) on female subjects, unless they have undergone a surgical procedure for sterilization or are post-menopausal (defined as more than 2 years have elapsed since their last menstruation in the absence of contraceptive use)
* A bone marrow aspirate with cytogenetics with or without biopsy with molecular testing.

Study Evaluations

Baseline Assessment

Patient testing will reflect the routine clinical operating practices of the Ottawa Hospital Blood and Marrow Transplant and Radiation Oncology Programs. The following measures and tests will be used to evaluate the status of the leukemia prior to treatment and the patient's pre-treatment organ function. They will be performed within 2 weeks of the first fraction of ED-TBI .

* History, physical examination, height and weight upon admission
* Urinalysis
* ECOG performance status
* HCT-specific cd-morbidity index
* CBC, differential
* Serum Creatinine, bilirubin, AST, ALT, ALP.
* INR, PTT, fibrinogen
* TSH
* A bone marrow aspirate with cytogenetics and molecular testing, with or without biopsy.

Post-transplant Assessments

Patient testing in the immediate period during ED-TBI and following alloHSCT will reflect the clinical operating practices of the Ottawa Hospital Blood and Marrow Transplant Program. The tests will be used to evaluate the severity of acute radiation toxicity, the time to engraftment, GVHD etc.

* History and physical exam to assess GVHD and other morbidity weekly until Day 100 post-transplant, then at four months, six months, one year, 18 months and two years post-transplant.

  * Acute GVHD will be evaluated according to the grading system in appendix 8
  * Chronic GVHD will be evaluated according to the grading system in appendix 9
* CBC at least three times a week from Day 0 until ANC > 0.5 x 109/L for 3 consecutive measurements over 3 or more days. Thereafter CBC at least twice per week until Day 28, then preferably weekly until Day 100, then at 12 months, 18 months and two years post-transplant
* Creatinine, bilirubin, alkaline phosphatase, ALT, AST, twice a week until Day 28 and then preferably weekly until 12 weeks, then at four months, six months, one year, eighteen months and two years post-transplant.
* Tacrolimus levels will be measured at least once weekly until the drug is tapered off.
* Serum CMV-PCR weekly for at least 6 months.
* Bone marrow aspirate and biopsy at Day 100 ±30 days on all patients. Bone marrow aspirate and biopsy at 12 ±3 months post-transplant is recommended, but not required, for all patients.
* Treat-related toxicity (RRT) assessments will be conducted weekly until Day 100 and additional toxicity assessments will be conducted on Day 100, 180, 365 and 730 post-transplant using the CTCAE V.4.
* Weekly urinalysis until discharge and then at 6, 12, 18 and 24 months.

The following tests will be performed at 6 months following treatment and then annually until 2 years after the transplant

* Bone Mineral Density
* TSH
* Serum Testosterone (males)
* LENT-SOMA Radiation Toxicity Scale
* Pulmonary Function Tests (Flow Rates, Diffusion Capacity, Lung Volumes and O2 Saturation by oximetry.)

The following will be performed at any time to look for relapse, if indicated (i.e. drop in the platelet count below 100 x 109 cells/L or in the neutrophil count below 1 x 109 cells/L, circulating blasts >0%, unrelated to treatment) or if there is any other reason to suspect relapse.

-Bone marrow aspirate +/- biopsy

Other tests may be added and the frequency of the above test may be changed depending on the clinical scenario during the transplant.

The following summary statistics will be obtained at the time of discharge from the alloHSCT hospital admission:

* Weight at discharge
* Number of units of blood and platelets administered
* Number of febrile days (t>38oC)
* Documented Infections
* Maximum adverse events according to CTCAE v.4
* Days admitted to the BMT Day hospital unit
* Days admitted to the BMT Inpatient unit
* Days admitted to the ICU
* Length of Hospital admission

ELIGIBILITY:
Inclusion Criteria

* All subjects must meet all of the following criteria to be eligible for the study. These will be evaluated within the four weeks prior to enrolment.
* Subject must have primary refractory AML, secondary AML, relapsed AML or high risk MDS
* Primary refractory AML is defined as:

A blast count in the bone marrow of >5% or the presence of any amount of circulating blasts, in the peripheral blood, after 1 cycle of induction chemotherapy.

* Secondary AML is defined as:

AML, except acute promyelocytic leukemia, arising from any haematological disease or from the exposure to chemotherapy for another unrelated malignancy.

* Relapsed AML is defined as:

Relapse (>5% blasts in the marrow) after having achieved a CR, of any duration.

* High risk myelodysplasia is defined as:

Myelodysplastic syndrome as defined by the WHO criteria with an international prognostic score (IPSS) of intermediate-2 or high

* Subjects must have a score of ≥2 on the scoring system for hematopoietic stem-cell transplantation for acute leukemia in relapse or primary induction failure
* Subjects must meet institutional guidelines for an alloHSCT.
* Subjects must have a matched related or a well- or partially-matched unrelated donor, acceptable to institutional guidelines who can donate either peripheral blood or bone marrow hematopoietic stem cells.
* Subjects must be of age ≥18 and ≤60 years.
* Subjects must have an ECOG performance score of 0,1, or 2
* Subjects must have the ability to comply with the protocol visit schedule and other protocol requirements.

Exclusion Criteria

* Subjects who have a score of < 2 on the scoring system for hematopoietic stem-cell transplantation for acute leukemia in relapse or primary induction failure
* Subjects who previously received an autoHSCT or alloHSCT
* Subjects who have previously received radiation therapy
* Subjects with a prior nephrectomy or a known history of a single kidney.
* Subjects with HIV-seropositivity.
* Subjects with a recent history of alcohol or drug abuse.
* Pregnant or lactating female subjects.
* Subject whose only donor is an umbilical cord donor
* Subjects whose only donor is an unrelated mismatched donor, according the recently published CIBMTR criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year post allogenic transplant
  The primary objective of this study is to determine the progression-free survival at 1 year, post alloHSCT, after ED-TBI followed by an alloHSCT for patients with refractory AML

SECONDARY OUTCOMES:
Engraftment | Within 100 day post transplant
  The time to neutrophil and platelet engraftment following ED-TBI and alloHSCT
Morbidity/Mortality | day 30, day 100, day 180 post transplant
  * The day 30 morbidity (frequency, severity and affected organ function) of ED-TBI
  * The day 30 mortality associated with ED-TBI and alloHSCT.
  * The day 100 morbidity (frequency, severity and affected organ function) of ED-TBI
  * The day 100 mortality associated with ED-TBI and alloHSCT.
  * The late (> 6 month and >1 year) morbidity and mortality of ED-TBI/alloHSCT
Relapse | 5 years post transplant
  * Relapse rate after alloHSCT
  * The pattern of relapse (blood and marrow vs. extramedullary)
  * The overall survival
GVHD | day 30, day 100, 180, 365 and 730 post transplant
  Incidence and severity of acute and chronic GVHD

OTHER OUTCOMES:
Evaluation of Safety | day 30, day 100, 180, 365 and 730 post transplant
  All patients who receive at least one fraction of ED-TBI will be used in the safety analysis.
  * The incidence of adverse and serious adverse events will be tabulated by, severity and relationship to the treatment.
  * Adverse and serious adverse events will be monitored on an ongoing basis by the investigators.
  * Adverse events will be categorized using the CTCAE v.4. Adverse events will be summarized at the following intervals post stem cell transplant: day 30, day 100, 180, 365 and 730.
Evaluation of Efficacy | day 30, day 100, 180, 365 and 730 post transplant
  Objective data to determine CR rate, rate of relapse, time-to-progression and overall survival will be collected and reported.
Duration of Study | 2-3 years
  Approximately, 5 patients from our institution will be eligible per year. Additional patients from cooperating centers could, potentially, add another 5 patients/year. Therefore, the duration of accrual is expected to be between 2-3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Sabloff, Principal Investigator — The Ottawa Hospital - Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Ottawa Hospital Research Institute — http://www.ohri.ca/